CLINICAL TRIAL: NCT07316829
Title: TRAnscriptional Profile of Peripheral Blood Cells in Patient With Chronic Kidney and Lung Rejection: Correlation With Response to Extracorporeal Photo-aphereSiS: : Studio Osservazionale-ambispettico.
Brief Title: TRAnscriptional Profile of Peripheral Blood Cells in Patient With Chronic Kidney and Lung Rejection: Correlation With Response to Extracorporeal Photo-aphereSiS
Acronym: TRACKLESS
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Marilena Gregorini, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: TRACKLESS
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-08

CONDITIONS: Graft Rejection; Kidney Transplantation; Lung Transplantation; Antibody-Mediated Rejection; Chronic Disease; Bronchiolitis Obliterans; HLA Antibodies; Antibodies, Donor-Specific; Immune Tolerance
Keywords: Extracorporeal photoapheresis; Antibody-mediated chronic rejection; Donor-specific antibodies; Kidney transplantation; Lung transplantation; Chronic lung allograft dysfunction; Bronchiolitis obliterans syndrome; Gene expression profiling; Treatment response biomarkers; Regulatory T cells
MeSH Terms: conditions — Chronic Disease; Bronchiolitis Obliterans; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral blood samples collected for gene expression profiling and immunological analyses.

GROUPS / COHORTS (2):
- Kidney transplant recipients receiving ECP: Adult kidney transplant recipients with biopsy-proven antibody-mediated chronic rejection who receive extracorporeal photoapheresis (ECP) as part of their treatment. Patients will be followed longitudinally with measurements of renal function, proteinuria, donor-specific antibodies, and gene expression profiling at baseline, 6 months, and 12 months.
- Lung transplant recipients receiving ECP: Adult lung transplant recipients diagnosed with chronic lung allograft dysfunction (CLAD) who receive extracorporeal photoapheresis (ECP) as part of their treatment. Patients will be followed longitudinally with measurements of pulmonary function (FEV1), donor-specific antibodies, and gene expression profiling at baseline, 6 months, and 12 months.

SUMMARY:
With this project, the research team aims to identify the molecular pathways associated with the response to extracorporeal photonchemioapheresis (ECP) in kidney or lung transplant patients suffering from chronic rejection, by analyzing gene expression in samples of peripheral blood mononuclear cells.

DETAILED DESCRIPTION:
Antibody-mediated chronic rejection (AMCR) is the leading cause of kidney graft loss. On average, more than 50% of patients resume dialysis within two years of diagnosis. The prevalence of AMCR reported in the literature varies, reaching up to 30%. The causes of chronic humoral rejection are not yet fully understood; however, its mechanism is based on donor-specific antibodies (DSAs), which may appear in the patient's serum and play a critical role. It remains unclear whether different inflammatory stimuli and/or inadequate immunosuppression induce their formation.

AMCR-related damage develops insidiously and often progresses rapidly to end-stage renal failure, with the onset of nephrotic-range proteinuria. For several years, it has been possible to detect and monitor DSAs in patient serum using the Luminex technique (LSAB: Luminex single antigen beads), which offers extremely high sensitivity and specificity.

De novo DSAs (dnDSAs) have been reported in 12-19% of kidney transplant recipients, and in 63% of cases their presence is associated with histological features of chronic rejection, high levels of proteinuria, and a rapid decline in glomerular filtration rate (GFR). It has been estimated that the reduction in GFR is four times greater in patients with dnDSAs than in age-matched transplant recipients without dnDSAs. Some authors report that even low dnDSA levels (MFI < 1000) are predictive of poor outcomes. The unfavorable prognosis associated with dnDSAs appears to depend on their ability to fix complement (C1q, C4d, and C3d), which confers increased cytotoxicity.

The diagnostic criteria for AMCR, revised at the 2013 Banff meeting, are threefold: (i) morphological evidence of chronic rejection in tissue, (ii) evidence of antibody interaction with the vascular endothelium, and (iii) serum positivity for DSAs.

Currently, there is no effective therapy for chronic humoral rejection, and there is broad consensus within the scientific community that prevention-through optimal organ allocation and adequate immunosuppressive regimens-remains the only viable strategy. Most published studies describe small patient cohorts treated with steroids and/or rituximab (RTX), high-dose intravenous immunoglobulin (IVIG), plasmapheresis (PHP), and/or bortezomib (BTZ) in addition to standard therapy. None of these treatments has demonstrated proven efficacy, while an increased risk of infection has been consistently reported.

Extracorporeal photoapheresis (ECP) is currently used for the treatment of cutaneous lymphoma, graft-versus-host disease (GVHD), and chronic lung transplant rejection. Several studies have shown preservation of transplanted organ function. ECP is well tolerated, has no significant side effects, and has recently been included in treatment guidelines for GVHD refractory to other therapies. Clinical trials are currently underway to evaluate its efficacy in chronic pulmonary rejection (bronchiolitis obliterans syndrome, BOS), liver transplantation, and chronic GVHD.

In kidney transplantation, ECP has been reported in cases of acute antibody-mediated rejection, recurrent acute rejection, refractory acute rejection, and steroid-resistant acute rejection, both as adjunctive prophylaxis to standard immunosuppression and as therapy in patients diagnosed with chronic rejection. In our experience, ECP treatment administered to 11 kidney transplant recipients with biopsy-proven AMCR and stage 2-3 chronic kidney disease resulted in stabilization of estimated GFR and proteinuria over a three-year follow-up period. Concurrently, DSA levels were reduced and completely eliminated in 73% of patients. Furthermore, we demonstrated that the therapeutic efficacy of ECP was mediated by an increase in regulatory T cells (Treg) and a decrease in Th17 cells.

In lung transplantation, long-term graft survival is also significantly affected by the development of chronic rejection, known as chronic lung allograft dysfunction (CLAD). CLAD is defined as a persistent decline in lung function-particularly a reduction in FEV1 of at least 20% compared with post-transplant baseline-in the absence of other identifiable causes. Chronic rejection was previously identified exclusively with bronchiolitis obliterans syndrome (BOS), an irreversible obstructive defect. More recent studies have described an additional phenotype, restrictive allograft syndrome (RAS). Although no universally accepted definition of RAS exists, emerging evidence suggests that BOS and RAS differ in pathological features, pathogenesis, clinical course, and natural history.

At present, no randomized controlled trials have evaluated ECP in lung transplantation, and, as in kidney transplantation, the mechanisms underlying its effects in chronic lung rejection remain unclear. Two small studies have suggested a role for ECP in the expansion of peripheral regulatory T-cell clones, while a more recent study indicates that ECP may modulate B cells and DSA production. Finally, there are currently no data supporting the early identification of so-called "responders" to ECP therapy.

Therefore, based on current knowledge, despite the increasingly widespread use of this treatment in various clinical settings, the mechanisms underlying the efficacy of ECP are not yet fully understood, particularly in the field of transplantation

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Kidney transplant recipients with biopsy-proven AMCR
* Lung transplant recipients with CLAD, defined as a persistent decline in FEV1 ≥ 20% compared with post-transplant baseline in the absence of other causes
* Patients receiving standard immunosuppressive therapy and eligible for Extracorporeal Photoapheresis (ECP)
* Ability to provide informed consent

Exclusion Criteria:

* Active infection or uncontrolled comorbidities that contraindicate ECP
* Pregnancy or breastfeeding
* Participation in another interventional trial that could interfere with outcomes
* Inability to comply with study procedures

Additional Notes:

* Both prevalent and incident cases may be included (ambispective design).
* Patients will be followed longitudinally for clinical outcomes, donor-specific antibodies, and gene expression profiling at baseline, 6 months, and 12 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes adult kidney and lung transplant recipients diagnosed with chronic antibody-mediated rejection (AMCR) or chronic lung allograft dysfunction (CLAD), respectively.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
omparison of gene expression profiles between responders and non-responders to Extracorporeal Photoapheresis (ECP) | 6 months (lung transplant cohort) and 12 months (kidney transplant cohort)
  The primary outcome is the difference in gene expression profiles between patients who respond and those who do not respond to ECP treatment. Response is defined based on stabilization or improvement of graft function (eGFR in kidney recipients, FEV1 in lung recipients) and reduction or elimination of donor-specific antibodies. Gene expression profiling will be performed on peripheral blood samples collected at baseline (T0) and after 6 months (lung) or 12 months (kidney) of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy